CLINICAL TRIAL: NCT03424642
Title: Interactive Ultrasound Examination as Psychological Support for Pregnant Women
Brief Title: Interactive Ultrasound Examination
Acronym: 4D ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 150613090915
Record Dates: First submitted 2018-01-05; First posted 2018-02-07 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Prenatal Anxiety
Keywords: prenatal depression; prenatal anxiety; prenatal mental disorders; interactive ultrasound examination; maternal-fetal relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive 4D-ultrasound examination (Experimental): Pregnant women who are randomized to 4D-ultrasound intervention group will receive additional 4D-ultrasound examinations 2-3 times between gestational weeks 25-32. Patients in this group will also receive psychologist's interview twice and fill out questionaries.
  Interventions: Behavioral: Interactive 4D-ultrasound examination
- Control group (No Intervention): Pregnant women who are randomized to control group will receive psychologist's interview twice twice and fill out questionaires.

INTERVENTIONS:
Behavioral: Interactive 4D-ultrasound examination — Randomized controlled trial
  Arms: Interactive 4D-ultrasound examination

SUMMARY:
Relationship between mother and child starts to develop during pregnancy and continues after birth. Drug abuse, depression, very young or old age, weak social network, mothers´ own negative experiences from childhood's relationships and fear of birth may weaken the normal development of maternal-fetal bonding during pregnancy. Gestational weeks 24-32 are crucial in the point of maternal-fetal bonding. Ultrasound examinations during pregnancy have shown to strengthen the early relationship between mother and fetus in every trimester, to diminish mother's anxiety, to improve mothers bonding to child and to guide mother towards healthier lifestyle. Mental images awaken emotional relationship to the child. It is possible to prevent the interference of the gestational process of forming mental images and to diminish the negative effects of gestational stress to the child by intervention, that further prevents the problems of the baby's first year. Psychological intervention, that supports the interaction between mother and child, combined to gestational ultrasound examination has not investigated before in pregnant women with risk to preterm birth, depressive symptoms or other mental symptoms.

DETAILED DESCRIPTION:
Relationship between mother and child starts to develop during pregnancy and continues after birth. The basis to it consists of mental images of self and spouse and observations of the baby via ultrasound examinations and sensations of the baby's movements. Drug abuse, depression, very young or old age, weak social network, mother's own negative experiences from childhood's relationships or fear of birth may weaken the normal development of maternal-fetal attachment. Gestational weeks between 24-32 are crucial in the point of maternal-fetal bonding. Preterm birth interrupts the development of the attachment. Studies have approved that parents' psychiatric morbidity predisposes the offspring to developmental and psychological problems. It's known that parents' depression predisposes their children to behavioral- and emotional disorders.

Prenatal depression leads to postnatal depression after birth in about 10 % of pregnant women. Depressive symptoms can reflect to expectancy and to emotions towards the unborn child and affect the quality of the early interaction between mother and baby. Mothers' depressive symptoms have link to pregnancy complications and to preterm birth. Anxiety and depression during the third trimester increases the risk to preterm birth. Anxiety during pregnancy has a connection to pre-eclampsia. The problems in maternal- fetal relationship originate from pregnancy and that's why timing treatment pregnancy is important. Pregnancy is opportune time to treat mothers' physical and psychic problems because the worry about the fetus motivates.

Gestational ultrasound has shown to strengthen the bonding towards the fetus in every trimester, to diminish mothers' anxiety, to improve mothers attachment to the fetus and to guide mother towards healthier lifestyle. Psychologic intervention combined with gestational ultrasound examination has detected to strengthen the maternal-fetal interaction in depressive mothers. Mental images awaken emotional bond to the unborn child. It is possible to prevent the disturbance of the process of forming mental images and to decrease the negative impact of gestational stress with gestational ultrasound examination. Interactive ultrasound examination has not explored before in pregnant women with risk to preterm birth, depressive and other mental symptoms. By awakening and strengthening mother's mental images of fetus decreases anxiety and other psychic symptoms.

The aim of the study is to develop a documented treatment model in specialist medical care to pregnant women who suffer from mental disorders in order to strengthen the early bonding via interactive ultrasound examination. The aim of the study is to find out if the interactive ultrasound examination improves interaction between mother and baby and does it improve baby's prognosis. To find out does the interactive ultrasound improve gestational bonding to fetus. To find out does the interactive ultrasound examination diminish mother's depressive and anguish symptoms. To find out the cost co efficiency in health care visits.

Pilot study was carried out with pregnant women who are hospitalized because of risk to preterm birth. 4D-ultrasound is done once and psychologist's interview after the examination. The aim of the pilot study was to map mothers' experiences of interactive ultrasound examination and to map their needs to psychological support in addition to interactive ultrasound examination before the actual randomized trial.

The research frame is controlled randomized trial. The sample size is 60 to both ultrasound intervention and to control group. The examinees are recruited from maternity clinics in Turku and surrounding cities. The main inclusion criteria are 10-14 points from EPDS-questionaire (Edinburgh pre/postnatal depression scale). EPDS is widely used questionaire in Finnish prenatal care in screening mental symptoms. Other inclusion criteria are singleton pregnancy, age over 18 years, fluent ability to speak Finnish and BMI under 35. Exclusion criteria are severe mental symptoms such as suicidality or psychotic symptoms. Depressive medication is not exclusive to this trial. All the participants will undergo psychologist's interview (WMCI, Working Model of The Child Interview) twice, the first interview will take place before randomization in gestational weeks 25 and the second on week 32. Examinees that end up in ultrasound intervention group will receive 2-3 4D-ultrasound examinations between gestational weeks 25-32. The focus of the 4D-ultrasound examination is to follow the fetus inside the womb and work on the mental images related to pregnancy and to the baby. The purpose is to hear the mother's thoughts and experiences about the fetus during the ultrasound examination. Doctor, who is familiar with gestational ultrasound examinations, tells under the examination what is seen and what the fetus does. It is possible to fetus' face and view its expressions with 4D-ultrasound. All the participants will answer to few questionairies: MAAS (Maternal Antenatal Attachment Scale),MPAS (Maternal Postnatal Attachment Scale), PRAQ-R2 (Pregnancy Related Anxiety Questionaire Revised) and SCL-90 (Symptoms checklist). Information regarding pregnancy and birth will be collected from medical records. The quality of mother-infant interaction will be observed 4 months postpartum with videotaped Parent-Child Early Relational Assessment- method.

Ethical committee of hospital district of southwest Finland has given approval to this study.

ELIGIBILITY:
Inclusion Criteria:

* pilot study(pregnant women who are hospitalized because of risk to preterm birth): singleton pregnancy, fluent in Finnish, age over 18
* randomized trial: EPDS 10-14 points, singleton pregnancy, fluent in Finnish, age over 18, BMI under 35

Exclusion Criteria:

* severe psychic symptoms e.g. suicidality, psychotic symptoms

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
prenatal depressive symptoms | Gestational weeks 21-24
  EPDS (Edinburgh Pre/Postnatal depression scale). 10 questions, scale 0-30 points, cut of for major depression is 15 points.
postnatal depressive symptoms | 4 months postpartum
  EPDS (Edinburgh Pre/Postnatal Depression Scale) 0-30 points, cut-off for major depression is 15 points.

SECONDARY OUTCOMES:
general anxiety | At gestational week 25 and at gestational week 32-33.
  SCL-90 (Symptom Checklist) measures general anxiety. Consists of 90 questions, each question contains 4 items. Higher score correlates positively with anxiety symptoms.
pregnancy related anxiety | At gestational week 25 and at gestational week 32-33
  PRAQ-R2 (Pregnancy Related Anxiety Questionaire Revised) Measures pregnancy related anxiety. Consists of 11 questions, each containing 5 items. Higher score correlates positively with pregnancy related anxiety.
maternal-fetal relations | At gestational week 25 and 32-33
  WMCI (Working Model of the Child Interview) is psychologists interview, that is a one-hour, semi-structured, exploring systematically the narrative patterns of parents' thoughts, feelings, and perceptions of their unborn baby and their emerging relationship. The scoring of the quality of parents' representations will be conducted from video recorded interviews. The quality and the content of the representations will be scored straight from the videotapes of the interviews using with the seven scales presented in the manual. The qualitative scales are richness of perceptions, openness to change, intensity of involvement, coherence, caregiving sensitivity, and acceptance. The content scales are infant difficulties and fear for the infant's safety. These scales will be scored with a Likert type scale ranging from 1 to 5. The parental representations will be classified based on the manual into three categories: balanced, disengaged, and distorted.
maternal-fetal attachment | At gestational week 25 and 32-33.
  MAAS (Maternal Antenatal Attachment Scale) is 19 questions containing questionaire. which focus on feelings, attitudes and behaviours towards the fetus with responses recorded on a 5 point Likert Scale. Maximum score is 95 points. High score correlates to strong attachment, low score to weak attachment.
maternal-fetal attachment | 4 months postpartum.
  MPAS (Maternal Postnatal Attachment Scale) is 19 questions containing questionaire. which focus on feelings, attitudes and behaviours towards the foetus with responses recorded on a 5 point Likert Scale. Maximum score is 95 points. High score correlates to strong attachment, low score to weak attachment.
maternal-fetal fetal relations | 4 months postpartum.
  Parent Child Early Relational Assessment (PCERA) observation. Videotaped interplay is analysed by psychologist.
  the foetus with responses recorded on a 5 point Likert Scale. Maximum score is 95 points. High score correlates to strong attachment, low score to weak attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Eeva MK Ekholm, ph d, Principal Investigator — TYKS
Locations (1):
- TYKS Naistenklinikka, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pulliainen H, Sari-Ahlqvist-Bjorkroth, Ekholm E. Does interactive ultrasound intervention relieve minor depressive symptoms and increase maternal attachment in pregnancy? A protocol for a randomized controlled trial. Trials. 2022 Apr 15;23(1):313. doi: 10.1186/s13063-022-06262-4. PMID 35428357